CLINICAL TRIAL: NCT04878770
Title: Use of the NMF Biomarker as Predictive Diagnostic for Effective Use of Cyclosporine and Dupilumab in the Treatment of Atopic Dermatitis
Brief Title: NMF-CsA-Dupi Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Suzanne G.M.A. Pasmans, Prof. S.G.M.A. Pasmans, MD PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC-2019-0568; 2019-003247-30 (EudraCT Number)
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Dermatitis, Atopic
Keywords: natural moisturizing factor; systemic treatment
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Adrenal Cortex Hormones; Cyclosporine; dupilumab

STUDY DESIGN:
Intervention Model Description: This is a partially-blinded randomized controlled trial that investigates if NMF-biomarker status has an effect on the effectiveness of systemic treatment with CsA in children with moderate-to-severe AD. It also investigates whether stratification on the NMF biomarker results in an improvement of efficiency in the use of systemic treatment with CsA in the treatment of moderate-to-severe AD.
Who Masked: Outcomes Assessor
Masking Description: Personnel involved assessing disease severity are blinded for the NMF biomarker result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical corticosteroids (control) (Active Comparator): This group will receive topical corticosteroids.
  Interventions: Drug: Topical corticosteroids
- Systemic cyclosporine (Active Comparator): This group will receive topical corticosteroids and systemic cyclosporin.
  Interventions: Drug: Topical corticosteroids; Drug: Systemic cyclosporine
- Systemic dupilumab (Active Comparator): his group will receive topical corticosteroids and systemic dupilumab.
  Interventions: Drug: Topical corticosteroids; Drug: Systemic dupilumab

INTERVENTIONS:
Drug: Topical corticosteroids — Topical corticosteroids (TCS) are registered for patients of all ages, and are together with emollients, the pillars in the basic treatment of atopic dermatitis. In this study, patients in both the intervention groups and control group are treated with daily emollients and a TCS of moderate to high potency if needed. Rescue medication with TCS of higher potency may be prescribed if basic therapy is inadequate in controlling AD symptoms.
Drug: Systemic cyclosporine — Systemic cyclosporine A (CsA) is an immunosuppressive therapy and is a registered treatment for AD in adults. According to national guidelines, CsA is the first choice for systemic treatment in children with moderate-to-severe AD.
  For CsA a starting dose of 4-5mg/kg/day is administered orally and then tapered down to 2-3mg/kg/day depending on clinical effect. Two doses will be taken at two fixed times per day. Treatment with systemic CsA will be continued for a total of 6 months.
  Other Names: Neoral
  Arms: Systemic cyclosporine
Drug: Systemic dupilumab — Dupilumab (DUPIXENT) is indicated for the treatment of children of 6 years and older with moderate-to-sever atopic dermatitis whos disease is not adequately controlled with topical prescription therapies or when those therapies are not advisable. DUPIXENT can be used with or without topical corticosteroids. rm: Active Comparator: Systemic dupilumab Dupilumab (DUPIXENT) is administered as a solution by subdermal injection according to national guidelines, based on age and body weight.
  Other Names: DUPIXENT
  Arms: Systemic dupilumab

SUMMARY:
The goal of this study is to investigate whether stratification of children with atopic dermatitis on the NMF biomarkers results in an improvement of effectiveness and efficiency in the use of systemic treatment (ciclosporin and dupilumab) in moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents, aged 2-18 years, with moderate-to-severe atopic dermatitis (diagnosed according to the UK working party criteria)
* Patient and parents/guardians able to participate in the study and willing to give written informed consent
* EASI (Eczema Area Severity Index) ≥ 6 at screening and baseline (corresponding with moderate-to-severe disease)
* IGA (Investigator Global Assessment) ≥ 3 at screening and baseline (corresponding with moderate-to-severe disease)

Exclusion Criteria:

* Children under the age of 2 years and patients older than 18 years
* Contraindication for ciclosporin
* Contraindication for dupilumab
* Patient (or one of the parents/guardians) not willing to be randomized
* Children with a history of any known primary immunodeficiency disorder
* Children with a history of cancer
* EASI < 6 at screening or baseline
* IGA < 3 at screening or baseline

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
EASI | t = 0, 1 month, 2 months, 3 months and 6 months
  Change from baseline Eczema Area and Severity Index (0-72) over the course of 6 months, with higher scores meaning worse outcomes.

SECONDARY OUTCOMES:
EASI75 | t = 1 month, 2 months, 3 months and 6 months
  Relative reduction of 75% from baseline EASI without the use of rescue medication
IGA 0 or IGA 1 | t = 0, 1 month, 2 months, 3 months and 6 months
  Proportion of patients that achieved IGA 0 or IGA 1 (Investigator's Global Assessment) without the use of rescue medication.
NRS-11 reduction for itch ≥ 4 points | t = 0, 1 month, 2 months, 3 months and 6 months
  Proportion of patients that achieved a reduction ≥4 points on the Numeric Rating Scale-11 (0-10) for itch intensity.
POEM | t = 0, 1 month, 2 months, 3 months and 6 months
  Change from baseline in Patient-Oriented Eczema Measure questionnaire (0-28) over the course of 6 months, with higher scores meaning worse outcomes.
SCORAD | t = 0, 1 month, 2 months, 3 months and 6 months
  Change from baseline in Scoring Atopic Dermatitis scale (0-103) over the course of 6 months, with higher scores meaning worse outcomes.
RECAP | t = 0, 1 month, 2 months, 3 months and 6 months
  Change from baseline in the Recap of Atopic Eczema questionnaire (0-28) over the course of 6 months, with higher scores meaning worse outcomes.

OTHER OUTCOMES:
CDLQI ≥4 years | t = 0, 3 months and 6 months
  Children's Dermatology Life Quality Index, in the context of a cost-effectiveness analysis
IDQoL <4 years | t = 0, 3 months and 6 months
  Infants' Dermatitis Quality of Life Index, in the context of a cost-effectiveness analysis
Emollients and steroid use in frequency and tubes used | t = 0, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months
  In context of a cost-effectiveness analysis: To assess the use of topical medication, including emollients, expressed in number of grams and/or used tubes, and changes therein during systemic treatment.
Healthcare costs related to the treatment of AD | Over the course of 6 months
  In context of a cost-effectiveness analysis: To assess medical specialist care, hospitalization, medication, and other costs directly associated with the treatment and recurrence.
Adverse events | Over the course of 6 months
  Adverse events related to therapy as reported at any time during treatment by patient, custodian or investigator.
NMF measured via Raman spectroscopy | t = - 2 weeks, 0, 3 months and 6 months
  Natural Moisturizing Factor, to acquire more knowledge about external and internal factors that influence the NMF biomarker
Microbiome profile | t = 0, 3 months and 6 months
  To investigate differences in microbiome profiles between patients with normal vs low NMF, and to investigate changes from baseline in microbiome profile during treatment, periodic swabs of nose, lesional skin, non-lesional skin and faeces will be obtained from patients.
Humoral blood panel (systemic arms) | t = 0, 1 month, 3 months and 6 months
  Changes in IgE during systemic treatment over the course of 6 months.
Humoral blood panel (topical arm) | t = 0 and 6 months
  Changes in IgE during topical treatment over the course of 6 months.
Cellular blood panel (systemic arm) | t = 0, 1 month, 3 months and 6 months
  Changes in leucocyte differentiation during systemic treatment over the course of 6 months.
FLG null mutations | t = 0
  Genotyping on skin barrier proteins, to acquire more knowledge about external and internal factors that influence atopic dermatitis and the NMF biomarker
Activity of atopy | t = 0, 3 months and 6 months
  The activity of rhinoconjunctivitis, asthma and food allergy examined by a pediatric allergist and pediatric pulmonologist.
Psychosocial factors (CBCL) | t = 0
  To investigate the influence of psychosocial factors in the patient on pediatric atopic dermatitis as assessed by the CBCL (Child Behaviour Checklist). Patients are assessed by questions grouped in empirically based syndrome scales: Aggressive Behavior, Anxious/Depressed, Attention Problems, Rule-Breaking Behavior, Somatic Complaints, Social Problems, Thought Problems, Withdrawn/Depressed. Higher percentile scores per scale indicate worse outcomes.
Psychosocial factors (OBVL) | t = 0
  To investigate the influence of psychosocial factors in the family on pediatric atopic dermatitis as assessed by the OBVL (OpvoedingsBelastingVragenLijst / Parenting Stress Questionnaire), with higher percentile scores indicating worse outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC - Sophia Children's Hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No